CLINICAL TRIAL: NCT06815055
Title: PREduKiné State of Play of Physiotherapy in the Postoperative Management of Prostate Cancer : Prospective, Monocentric, National Survey, Aiming to Explore the Technics of Physiotherapy
Brief Title: State of Play of Physiotherapy in the Postoperative Management of Prostate Cancer : Prospective, Monocentric, National Survey, Aiming to Explore the Technics of Physiotherapy (PREduKiné)
Acronym: PREduKiné
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Roubaix (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-010
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Radical Prostatectomies; Rehabilitation Outcome; Prostate Cancer; Prostate Cancer Surgery; Rehabilitation Exercise
Keywords: radical prostatectomy; rehabilitation; continence; quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Quality of life questionnary — Subjects will be call 1 month and 6 months after prostetectomy to evaluate the type of reeducation received and they will be evaluated with the help of QoL questionnaries : KHQ-HR QoL and ICIQ-SF QoL

SUMMARY:
In France, a considerable number of radical prostactectomy for cancer is carried out every year.This number was estimated at 20.000 in 2016.This surgery may have negative impact on the continence's subjects and their quality of life. The rehabilitation, preoperative or postoperative, practiced by a physiotherapist, can reduced those side effects. The rehabilitation techniques are many and their efficacy may differ.

No study where found about the clasification and evaluation of those rehabilitation techniques.

DETAILED DESCRIPTION:
Investigator aim to create homogeneous clusters of subjects according to the rehabilitation techniques they have received during the preoperative or postoperative period, using a survey replied 6 months after the surgery.

To achieve that goal, invesgator will call subjects conduct two interviews. The first interview will take place around one month after the radical prostatectomy and the second around 6 month after the surgery.

During those interviews, investigator will question subjects about the rehabilitation techniques practiced on them, about their continence and quality of life. To evaluate the continence investigator will use the survey ICIQ-SF. To evaluate the quality of life, investagator will use the survey KHQ-HR Qol.

ELIGIBILITY:
Inclusion Criteria:

* men who has undergone a radical prostactectomy to treat a prostatic adenocarcinoma
* having a follow up postoperative consultation between one and two month after the surgery
* being able to answer to respond the questions during the interviews
* agreeing to participate by signing informed consent form

Exclusion Criteria:

* undergoing an adjuvant therapy as radiotherpy, chemotherapy and hormone therapy
* Refusing to take part in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population concerned by the study is national french territory. Subjects must have an postoperative follow up performing by an urologist.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Set up homogeneous groups of subjects (clusters) | It will take place around six months after the surgery.
  The primary outcome is a survey questionning the subject about the rehabilitation techniques realised during the post operative period. This survey will be asked during a phone interview directed by investgator.